CLINICAL TRIAL: NCT05918913
Title: Expanded Access Program for SNDX-5613 in Patients With Relapsed/Refractory Acute Leukemias With Genetic Alterations Associated With HOXA Overexpression
Brief Title: Expanded Access Program for Revumenib
Status: No longer available | Type: Expanded Access
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNDX-5613-0707
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Acute Leukemia
Keywords: SNDX-5613; Acute Leukemia; Refractory leukemia; Relapsed leukemia; KMT2A; NPM1; UBTF tandem duplication; Revumenib; Revuforj
MeSH Terms: conditions — Recurrence; Leukemia | interventions — revumenib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Revumenib — Revumenib administered orally every 12 hours.
  Other Names: SNDX-5613; Revuforj

SUMMARY:
This expanded access program will provide an investigational treatment option in a controlled clinical setting for participants who are not otherwise eligible to participate in other Syndax-sponsored clinical studies and have no approved treatment options.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participant aged ≥6 months.
* Not eligible for participation in an ongoing clinical study and have no approved treatment options.
* Participant or participant's health care proxy is able and willing to provide written informed consent and able to follow study instructions.
* Relapsed or refractory (R/R) acute leukemia, as defined by standardized criteria, after standard of care therapy, including but not limited to 1 or 2 cycles of intensive chemotherapy, or venetoclax combinations:

  1. R/R leukemia is defined by the presence of ≥5% blasts in the bone marrow and/or persistence or reappearance of peripheral blasts.
  2. Participants with persistent leukemia after initial therapy or recurrence of leukemia at any time after achieving a response during or after the course of treatment (including allogeneic hematopoietic stem cell transplant [HSCT]) are eligible.
  3. Participants with isolated extra-medullary disease are allowed if extramedullary disease was confirmed with biopsy.
  4. Participants previously treated on a revumenib clinical study who are entering the expanded access program for post-transplant maintenance because they are not eligible to receive revumenib on study or because the study is closed are not required to meet the R/R status.
  5. Participants who underwent HSCT and are eligible to resume treatment with revumenib will be dosed with the last revumenib tolerated dose before transplant.
* Acute leukemia harboring a lysine (K) methyltransferase 2A gene rearrangement (KMT2Ar), nucleoporin 98 rearrangement, nucleophosmin 1 mutation (or mutated) or any other genetic alteration with overexpression of HOXA genes predicted to potentially respond to menin inhibitors.

  * Note: As revumenib is now approved in the United States, only participants with a KMT2Ar who are not included in the United States prescribing information indication or cannot be accurately dosed (within a 20% margin) with commercial supply and require use of oral solution will be allowed into the study.
* Adequate liver, renal, and cardiac function.
* Use of highly effective methods of contraception are required for females and males of childbearing potential from the time of enrollment through 120 days following the last study intervention dose.

For participants currently being treated with revumenib in a Syndax-sponsored clinical study or Syndax investigator-sponsored trial, the following criteria must be met:

* In the opinion of the Investigator, participant demonstrated acceptable benefit from and tolerability of the study intervention.
* Participant is considered compliant with study intervention and procedures.
* Participant does not meet any criteria for study intervention discontinuation.
* Investigator and participant agree to continue study intervention treatment.
* Participant continues to experience clinical benefit.

Key Exclusion Criteria:

* Evidence of uncontrolled infection.
* Pregnant or nursing women.
* Cardiac or gastrointestinal disease.
* Graft-Versus-Host Disease (GVHD): Signs or symptoms of acute or chronic GVHD >Grade 1 within 4 weeks of enrollment. All transplant participants must have been off all systemic immunosuppressive therapy and calcineurin inhibitors for at least 1 week before enrollment, with the exception of steroids.
* History of or any concurrent condition, therapy, laboratory abnormality, or allergy to excipients that, in the Investigator's opinion, either may interfere with the participant's participation or results in the conclusion that it is not in the best interest of the participant to participate.
* Participants receiving other antileukemic therapy within 14 days of start of study drug and who have not recovered from previous adverse reactions.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Syndax Pharmaceuticals
Locations (35):
- United States (35):
  - Alabama Center for Childhood Cancer And Blood Disorders, Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - City of Hope at Orange County Lennar Foundation Cancer Center, Irvine, California
  - UCLA, UCLA RRMC, Drug Information Center, Department of Pharmaceutical Services Drug Supply Shipment, Los Angeles, California
  - Lucile Packard Children's Hospital-Stanford, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Center for Cancer and Blood Disorders, Colorado Children's Hospital, Aurora, Colorado
  - HCTU, Division of Hematology, University of Colorado, Anschutz Medical Center, Aurora, Colorado
  - Advent Health Orlando, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospital, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts
  - Children's Mercy Hospital-Kansas City, Kansas City, Missouri
  - Siteman Cancer Center - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, Long Island City, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Division of Hematology and Oncology, Division of Pulmonary, Critical Care and Sleep Medicine, Vontz Center for Molecular Studies, Cincinnati, Ohio
  - OSU Medical Center, Columbus, Ohio
  - Doernbecher Children's Hospital, Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Memorial Hermann-Texas Medical Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Division of Hematology and Hematologic Malignancies, University of Utah-Huntsman Cancer Hospital, Salt Lake City, Utah
  - Seattle Children's Research Institute, Seattle Childrens Hospital, Seattle, Washington